CLINICAL TRIAL: NCT02294058
Title: A Phase 3, Multi-Center, Randomized, Double-Blind, Double-Dummy, Active Controlled, Parallel Group Study To Evaluate The Efficacy And Safety Of RPC1063 Administered Orally To Relapsing Multiple Sclerosis Patients
Brief Title: Study of Ozanimod (RPC1063) in Relapsing Multiple Sclerosis (MS)
Acronym: SUNBEAM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RPC01-301; 2014-002320-27 (EudraCT Number)
Record Dates: First submitted 2014-08-05; First posted 2014-11-19 (Estimated); Results first posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Multiple Sclerosis
Keywords: MS; RMS; Multiple Sclerosis; Relapsing Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — ozanimod; Interferon beta-1a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Interferon beta-1a (Active Comparator): Participants received 30 µg interferon beta-1a by intramuscular (IM) injection weekly and matching placebo capsules (identical in physical appearance to ozanimod) orally once a day until the last participant had been treated for 12 months.
  Interventions: Drug: Interferon beta-1a; Drug: Placebo to ozanimod
- Ozanimod 0.5 mg (Experimental): Participants received ozanimod 0.5 mg capsules orally once a day and an intramuscular placebo injection (identical in appearance to Interferon) weekly until the last participant had been treated for 12 months.
  Interventions: Drug: Ozanimod; Drug: Placebo to interferon beta-1a
- Ozanimod 1 mg (Experimental): Participants received ozanimod 1 mg capsules orally once a day and an intramuscular placebo injection (identical in appearance to Interferon) weekly until the last participant had been treated for 12 months.
  Interventions: Drug: Ozanimod; Drug: Placebo to interferon beta-1a

INTERVENTIONS:
Drug: Ozanimod — Capsules for oral administration once a day
  Other Names: RPC1063; Zeposia®
  Arms: Ozanimod 0.5 mg; Ozanimod 1 mg
Drug: Interferon beta-1a — Administered by intramuscular injection once a week
  Other Names: Avonex®; IFN β-1a
  Arms: Interferon beta-1a
Drug: Placebo to ozanimod — Matching placebo capsules administered orally once a day
  Arms: Interferon beta-1a
Drug: Placebo to interferon beta-1a — Placebo intramuscular injection once a week
  Arms: Ozanimod 0.5 mg; Ozanimod 1 mg

SUMMARY:
The purpose of this study is to determine whether ozanimod is effective in the treatment of relapsing multiple sclerosis (RMS).

ELIGIBILITY:
Inclusion Criteria:

* Multiple sclerosis as diagnosed by the revised 2010 McDonald criteria
* EDSS score between 0 and 5.0 at baseline

Exclusion Criteria:

• Primary progressive multiple sclerosis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1346 (Actual)
Dates: Start 2014-12-03 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2016-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Sheffiled, MD, Study Director — Celgene
Locations (224):
- United States (40):
  - Xenosciences Inc, Phoenix, Arizona
  - St Josephs Hospital and Medical Center, Phoenix, Arizona
  - Northwest Neuro Specialists PLLC, Tucson, Arizona
  - Alta Bates Summit Medical Center, Berkeley, California
  - Collaborative Neuroscience Network Inc, Long Beach, California
  - University of California Davis Medical Center, Sacramento, California
  - Multiple Sclerosis Center at UCSF, San Francisco, California
  - Denver Neurological Clinic, Denver, Colorado
  - Neurology Associates PA, Maitland, Florida
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - Infinity Clinical Research LLC, Pompano Beach, Florida
  - Neurostudies Inc, Port Charlotte, Florida
  - Roskamp Institute, Sarasota, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - Meridien Research, Tampa, Florida
  - West Georgia Sleep Disorder Center and Neurology Associates, Douglasville, Georgia
  - Consultants In Neurology, Northbrook, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - MidAmerica Neuroscience Research Foundation, Lenexa, Kansas
  - Associates In Neurology, Lexington, Kentucky
  - Norton Healthcare, Louisville, Kentucky
  - Henry Ford Health System, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Minneapolis Clinic of Neurology, Golden Valley, Minnesota
  - Washington University, St Louis, Missouri
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - Neurology Specialists of Monmouth County PA, West Long Branch, New Jersey
  - Neuro Medical Care Associates PLLC, Johnson City, New York
  - Raleigh Neurology Associates PA, Raleigh, North Carolina
  - Neurology and Neuroscience Associates Inc., Akron, Ohio
  - Neurological Research Institute Inc, Columbus, Ohio
  - Providence Multiple Sclerosis Center, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Hope Neurology MS Center, Knoxville, Tennessee
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Bhupesh Dihenia MD PA, Lubbock, Texas
  - EvergreenHealth, Kirkland, Washington
  - The Polyclinic, Seattle, Washington
  - Neurology of Neurosurgery Associates of Tacoma, Tacoma, Washington
  - Center for Neurological Disorders, Milwaukee, Wisconsin
- Belarus (6):
  - Grodno Clinical Regional Hospital, Grodno
  - Minsk Municipal Clinical Hospital 5, Minsk
  - Republican Scientific and Practical Centre of Neurology and Neurosurgery, Minsk
  - Minsk City Clinical Hospital 9, Minsk
  - Vitebsk Regional Diagnostic Centre, Vitebsk
  - Vitebsk Regional Clinical Hospital, Vitebsk
- Bosnia and Herzegovina (3):
  - Clinical Center Banja Luka, Banja Luka
  - Clinical Center University of Sarajevo, Sarajevo
  - University Clinical Center Tuzla, Tuzla
- Bulgaria (9):
  - Military Medical Academy HBAT, Pleven
  - Multiprofile Hospital for Active Treatment of Neurology and Psychiatry Sv Naum EAD, Sofia
  - Multiprofile Hospital for Active Treatment National Cardiology Hospital EAD, Sofia
  - Multiprofile Hospital for Active Treatment Tokuda Hospital Sofia, Sofia
  - University Multiprofile Hospital for Active Treatment Aleksandrovska EAD, Sofia
  - University Multiprofile Hospital for Active Treatment Sveti Ivan Rilski EAD, Sofia
  - University Multiprofile Hospital for Active Treatment Tsaritsa Yoanna ISUL EAD, Sofia
  - Military Medical Academy - MHAT, Sofia
  - Multiprofile Hospital for Active Treatment Sveta Marina EAD, Varna
- Clinique Neuro Outaouais, Gatineau, Quebec, Canada
- Croatia (6):
  - Clinical Hospital Osijek, Osijek
  - General Hospital Varazdin, Varaždin
  - Clinical Hospital Center Zagreb, Zagreb
  - Clinical Hospital Dubrava, Zagreb
  - Clinical Hospital Sestre Milosrdnice, Zagreb
  - Clinical Hospital Sveti duh, Zagreb
- Czechia (8):
  - University Hospital Brno, Brno
  - Fakultni nemocnice u sv Anny v Brne, Brno
  - Private Neurological Practice Radomir Talab MD, Hradec Králové
  - University Hospital Hradec Kralove, Hradec Králové
  - Nemocnice Jihlava prispevkova organizace, Jihlava
  - Fakultni Nemocnice Olomouc, Olomouc
  - Vseobecna Fakultni Nemocnice v Praze, Prague
  - Krajska zdravotni as Nemocnice Teplice oz, Teplice
- Estonia (3):
  - East Tallinn Central Hospital, Tallinn
  - West Tallinn Central Hospital, Tallinn
  - Tartu University Hospital, Tartu
- Georgia (6):
  - Aversi Clinic LTD, Tbilisi
  - Khechinashvili University Hospital, Tbilisi
  - LTD MediClubGeorgia, Tbilisi
  - Sarajishvili Institute of Neurology, Tbilisi
  - Curatio JSC, Tbilisi
  - Ltd DEKA, Tbilisi
- Germany (12):
  - Praxis Dr. Wilfried Luer, Berlin
  - St. Joseph Krankenhaus Berlin, Berlin
  - Asklepios Fachklinikum Teupitz, Brandenburg
  - DataMed GmbH, Cologne
  - Universitatsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - Heinrich Heine Universitat Dusseldorf, Düsseldorf
  - Universitatsklinikum Leipzig, Leipzig
  - Klinikum der Stadt Ludwigshafen gGmbH, Ludwigshafen am Rhein
  - Klinikum der Philipps Universitat Marburg, Marburg
  - St. Josefs-Krankenhaus Potsdam-Sanssouci GmbH, Potsdam
  - Krankenhaus der Barmherzigen Brueder, Trier
  - NeuroPoint Akademie, Ulm
- Hungary (2):
  - Kenezy Gyula Korhaz es Rendelointezet, Debrecen
  - Pest Megyei Flor Ferenc Korhaz, Kistarcsa
- Latvia (3):
  - Latvian Maritime Medicine Centre, Riga
  - Riga East Clinical University Hospital clinic Gailezers, Riga
  - Pauls Stradins Clinical University Hospital, Riga
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas
  - Klaipeda University Hospital, Klaipėda
- Moldova (3):
  - IMSP Institutul de Medicina Urgenta, Chisinau
  - Municipal Clinical Hospital Sf Arhanghel Mihail, Chisinau
  - Institutul de Neurologie si Neurochirurgie, Chisinau
- Zuyderland Medisch Centrum, Sittard-Geleen, Netherlands
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Waikato Hospital, Hamilton
- Poland (25):
  - B&B Robert Bonek, Pawel Bochniak, Spolka Cywilna, Bydgoszcz
  - Powiatowy Zespol Zakladow Opieki Zdrowotnej Szpital w Czeladzi, Czeladź
  - Copernicus Podmiot Leczniczy Sp. z o.o., Gdansk
  - Akson Clinical Research Maciejowski Bielecki Sp. Jawna, Jarosław
  - Niepubliczny Zaklad Opieki Zdrowotnej NEURO-MEDIC, Katowice
  - M.A.- Lek A.M.Maciejowscy Spolka Cywilna, Katowice
  - Novo-Med Zielinski i wsp. Sp.J., Katowice
  - NEURO- CARE Site Management Organization Gabriela Klodowska-Duda, Katowice
  - RESMEDICA Spolka z o.o., Kielce
  - Niepubliczny Zespol Leczniczo-Rehabilitacyjny Centrum Kompleksowej Rehabilitacji, Konstancin-Jeziorna
  - Centrum Neurologii Krzysztof Selmaj, Lódzkie
  - NZOZ NEUROMED M. I M. Nastaj Spolka Partnerska, Lublin
  - Wojewodzki Szpital Specjalistyczny im Stefana Kardynala Wyszynskiego, Lublin
  - Samodzielny Publiczny Centralny Szpital Kliniczny, Mazowieckie
  - Neurologiczny NZOZ Centrum Leczenia SM Osrodek Badan Klinicznych Dr n med Hanka Hertmanowska, Plewiska
  - Niepubliczny Zaklad Opieki Zdrowotnej KENDRON, Podlaskie
  - Indywidualna Specjalistyczna Praktyka Lekarska dr nmed Monika Lyczak, Pomorskie
  - Niepubliczny Zaklad Opieki Zdrowotnej NEUROKARD Ilkowski i Partnerzy Spolka Partnerska Lekarzy, Poznan
  - SPZOZ Wojewodzki Szpital Specjalistyczny nr 3 w Rybniku, Rybnik
  - Centrum Medyczne Medyk, Rzeszów
  - Indywidualna Specjalistyczna Praktyka Lekarska Zbigniew Cebulski, Warminsko-mazurskie
  - Szpital Czerniakowski Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Warsaw
  - Centrum Medyczne NeuroProtect, Warsaw
  - Instytut Psychiatrii i Neurologii, Warsaw
  - Centrum Medyczne doktorA, Warsaw
- Portugal (5):
  - Hospital Garcia de Orta, Almada
  - Hospital de Braga, Braga
  - Centro Hospitalar E Universitario de Coimbra EPE, Coimbra
  - Hospital Beatriz Angelo, Loures
  - Campus Neurologico Senior, Torres Vedras
- Romania (6):
  - Fundeni Clinical Institute, Bucharest
  - Colentina Clinical Hospital, Bucharest
  - Cluj Clinical County Hospital, Cluj-Napoca
  - Cai Ferate Clinical Hospital, Constanța
  - Sibiu Emergency County Clinical Hospital, Sibiu
  - Timisoara Emergency County Clinical Hospital, Timișoara
- Russia (39):
  - Arkhangelsk Regional Clinical Hospital, Arkhangelsk
  - Regional Clinical Hospital, Barnaul
  - Belgorod Regional Clinical Hospital, Belgorod
  - Bryansk Regional Hospital 1, Bryansk
  - Chelyabinsk City Clinical Hospital 3, Chelyabinsk
  - Research Medical Complex Vashe Zdorovie, Kazan'
  - Kemerovo Regional Clinical Hospital, Kemerovo
  - Regional Clinical Hospital, Khanty-Mansiysk
  - Kirov City Clinical Hospital 1, Kirov
  - Krasnoyarsk State Medical Academy, Krasnoyarsk
  - Kursk Regional Clinical Hospital, Kursk
  - Central Clinical Hospital 2 na NA Semashko OAO RZhD, Moscow
  - City Clinical Hospital 24, Moscow
  - City Clinical Hospital 1 na NIPirogov, Moscow
  - Research Center of Neurology of RAMS, Moscow
  - City Clinical Hospital 11, Moscow
  - Nizhniy Novgorod City Hospital 33, Nizhny Novgorod
  - City Clinical Hospital 3 Nizhniy Novgorod Geriatrics Centre, Nizhny Novgorod
  - Siberian Regional Medical Center, Novosibirsk
  - Novosibirsk State Medical University, Novosibirsk
  - Penza Regional Clinical Hospital na NN Burdenko, Penza
  - Perm State Medical Academy, Perm
  - Republican Hospital na VA Baranov, Petrozavodsk
  - Pyatigorsk City Hospital 2, Pyatigorsk
  - Rostov Regional Clinical Hospital, Rostov-on-Don
  - City Hospital 31, Saint Petersburg
  - City Hospital Nikolaevskaya Bolnitsa, Saint Petersburg
  - St. Petersburg Multi Field City Hospital 2, Saint Petersburg
  - First St Petersburg State Medical University na IP Pavlov, Saint Petersburg
  - Institute of Human Brain RAN, Saint Petersburg
  - City Clinical Hospital 40, Saint Petersburg
  - Samara Regional Clinical Hospital named after MI Kalinin, Samara
  - Smolensk State Medical Academy, Smolensk
  - Siberian State Medical University, Tomsk
  - Regional State Budget Institution of Healthcare Tver Regional Clinical Hospital, Tver'
  - Neftyanik Medical and Sanitary Unit, Tyumen
  - Kuvatov Republican Clinical Hospital, Ufa
  - Yaroslavl Clinical Hospital 8, Yaroslavl
  - Sverdlovsk Regional Clinical Hospital 1, Yekaterinburg
- Serbia (6):
  - Clinical Center of Serbia, Belgrade
  - Clinical Hospital Centar Zvezdara, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Hospital Centre Zemun, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - Clinical Center Nis, Niš
- Spain (5):
  - Hospital Universitario Vall D hebron, Barcelona
  - Hospital Arnau de Vilanova, Lleida
  - Complejo Hospitalario de Navarra, Pamplona/ Navarra
  - Hospital Moises Broggi, Sant Joan Despí
  - Hospital Clinico Universitario de Valencia, Valencia
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Karolinska Universitetssjukhuset Solna, Stockholm
- Ukraine (24):
  - MI Cherkasy Regional Hospital of Cherkasy Regional Council, Cherkasy
  - Hospital 4 of Chernihiv City Council, Chernihiv
  - Municipal Treatment and Preventive Institution Chernihiv Regional Clinical Hospital, Chernihiv
  - Municipal Institution Chernivtsi Regional Psychiatric Hospital, Chernivtsi
  - Municipal Institution Dnipropetrovsk Regional Clinical Hospital na I.I. Mechnykov, Dnipropetrovsk
  - Ivano Frankivsk City Clinical Hospital 1, Ivano-Frankivsk
  - Regional Clinical Hospital., Ivano-Frankivsk
  - State Treatment and Prevention Institution Central Clinical Hospital of Ukrzaliznytsya, Kharkiv
  - Regional Clinical Hospital Center for Emergency Medical Care and Disaster Medicine, Kharkiv
  - Municipal Institution of Health Care Kharkiv Clinical City Hospital 7, Kharkiv
  - National Research Center for Radiation Medicine, Institute of Clinical Radiology, Kyiv
  - Kyiv City Clinical Hospital 4, Kyiv
  - Volyn Regional Clinical Hospital, Lutsk
  - Lviv Regional Clinical Hospital, Lviv
  - Municipal City Clinical Hospital 5, Lviv
  - Center for Reconstructive and Rehabilitation Medicine University Clinic of ONMedU, Odesa
  - Municipal Institution Odesa Regional Clinical Hospital, Odesa
  - Regional Clinical Hospital na NV Sklifosovskyi, Poltava
  - Regional Clinical Center of Neurosurgery and Neurology, Uzhhorod
  - Municipal Institution Vinnytsia Regional Psychoneurological Hospital na OI Yushchenko, Vinnytsia
  - Municipal Institution City Clinical Hospital 2, Zaporizhya
  - Municipal Institution 6th City Clinical Hospital of Zaporizhzhia City Council, Zaporizhzhia
  - Municipal Institution Zaporizhzhia, Zaporizhzhia
  - Regional Clinical Hospital na OFHerbachevskyi of Zhytomyr Regional Council, Zhytomyr
- United Kingdom (4):
  - University Hospital of Wales, Cardiff
  - Raigmore Hospital, Inverness
  - Kings College Hospital, London
  - Royal Hallamshire Hospital Sheffield Teaching Hospitals NHS Trust, Sheffield

REFERENCES:
- [Background] Comi G, Kappos L, Selmaj KW, Bar-Or A, Arnold DL, Steinman L, Hartung HP, Montalban X, Kubala Havrdova E, Cree BAC, Sheffield JK, Minton N, Raghupathi K, Ding N, Cohen JA; SUNBEAM Study Investigators. Safety and efficacy of ozanimod versus interferon beta-1a in relapsing multiple sclerosis (SUNBEAM): a multicentre, randomised, minimum 12-month, phase 3 trial. Lancet Neurol. 2019 Nov;18(11):1009-1020. doi: 10.1016/S1474-4422(19)30239-X. Epub 2019 Sep 3. PMID 31492651
- [Result] Cree B, et al. The RADIANCE and SUNBEAM phase 3 studies of ozanimod in relapsing multiple sclerosis: study design and baseline characteristics. Presented at the 69th Annual American Academy of Neurology Meeting, April 22-28, 2017, Boston, MA. Abstract No. P6-344
- [Derived] Harris S, Comi G, Cree BAC, Arnold DL, Steinman L, Sheffield JK, Maddux R, Southworth H, Kappos L, Cohen JA. Glial Fibrillary Acidic Protein as a Marker of Disease in Relapsing Multiple Sclerosis: Post Hoc Analysis of Phase 3 Ozanimod Trials. Eur J Neurol. 2025 Jun;32(6):e70222. doi: 10.1111/ene.70222. PMID 40462564
- [Derived] DeLuca J, Schippling S, Montalban X, Kappos L, Cree BAC, Comi G, Arnold DL, Hartung HP, Sheffield JK, Liu H, Silva D, Cohen JA. Effect of Ozanimod on Symbol Digit Modalities Test Performance in Relapsing MS. Mult Scler Relat Disord. 2021 Feb;48:102673. doi: 10.1016/j.msard.2020.102673. Epub 2020 Dec 10. PMID 33454584

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 152 sites in 20 countries in Eastern and Western Europe, the United States, and New Zealand. Between December 2014 and November 2015, 1656 participants were screened, of whom 1346 were eligible and enrolled.
Pre-assignment Details: Participants were randomly assigned to one of three treatment groups in a 1:1:1 ratio. Randomization was stratified by Baseline Expanded Disability Status Scale (EDSS) score (≤ 3.5, > 3.5) and country.
Groups:
- Interferon Beta-1a: Participants received 30 µg interferon beta-1a (IFN β-1a) by intramuscular (IM) injection weekly and matching placebo capsules (identical in physical appearance to ozanimod) orally once a day until the last participant had been treated for at least 12 months.
- Ozanimod 0.5 mg: Participants received ozanimod 0.5 mg orally once a day and a placebo intramuscular injection (identical in appearance to Interferon) weekly until the last participant had been treated for at least 12 months.
- Ozanimod 1 mg: Participants received ozanimod 1 mg orally once a day and a placebo intramuscular injection (identical in appearance to Interferon) weekly until the last participant had been treated for at least 12 months.
Period: Overall Study
Arm/Group | Interferon Beta-1a | Ozanimod 0.5 mg | Ozanimod 1 mg
Started | 448 | 451 | 447
Safety Population (Three participants randomized to the interferon beta-1a group received ozanimod in error at some visits (2 participants received ozanimod 0.5 mg and 1 participant received ozanimod 1 mg) and are counted in the ozanimod groups in the Safety Population.) | 445 | 453 | 448
Completed | 412 | 425 | 418
Not Completed | 36 | 26 | 29
Not completed — Adverse Event | 16 | 7 | 13
Not completed — Lack of Efficacy | 3 | 3 | 0
Not completed — Lost to Follow-up | 1 | 0 | 2
Not completed — Withdrawal by Subject | 10 | 14 | 13
Not completed — Physician Decision | 2 | 1 | 0
Not completed — Miscellaneous | 4 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population consisted of all randomized participants who received at least 1 dose of study drug; participants were analyzed according to the treatment they were randomized to receive and not according to what they actually received, if different.
Groups:
- Interferon Beta-1a: Participants received 30 µg interferon beta-1a by IM injection weekly and matching placebo capsules orally once a day until the last participant had been treated for at least 12 months.
- Ozanimod 0.5 mg: Participants received ozanimod 0.5 mg orally once a day and a placebo intramuscular injection weekly until the last participant had been treated for at least 12 months.
- Ozanimod 1 mg: Participants received ozanimod 1 mg orally once a day and a placebo intramuscular injection weekly until the last participant had been treated for at least 12 months.
- Total: Total of all reporting groups
Arm/Group | Interferon Beta-1a | Ozanimod 0.5 mg | Ozanimod 1 mg | Total
Number analyzed (Participants) | 448 | 451 | 447 | 1346
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (9.11) | 36.0 (9.43) | 34.8 (9.24) | 35.6 (9.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 300 | 311 | 283 | 894
  Male | 148 | 140 | 164 | 452
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 0 | 2 | 0 | 2
  Asian | 0 | 1 | 1 | 2
  White | 447 | 447 | 446 | 1340
  Other | 1 | 1 | 0 | 2
Region [Count of Participants; unit: Participants] — Eastern Europe includes Belarus, Bosnia and Herzegovina, Bulgaria, Croatia, Estonia, Georgia, Latvia, Lithuania, Moldova, Poland, Romania, Russia, Serbia, and Ukraine.
  Rest of world includes the United States, Germany, Portugal, Spain, Sweden, and New Zealand.
  Participants
    Rest of World | 29 | 32 | 32 | 93
    Eastern Europe | 419 | 419 | 415 | 1253
Expanded Disability Status Scale (EDSS) [Mean (Standard Deviation); unit: units on a scale] — The EDSS is a scale for quantifying disability in MS. Eight functional systems (visual, brain stem, pyramidal, cerebellar, sensory, bowel & bladder, cerebral, and other functions) are scored on a scale of 0 (no disability) to 5 or 6 (more severe disability). Ambulation is also scored. Based on scores in these 8 functional systems and gait, an overall score ranging from 0 (normal) to 10 (death due to MS) in 0.5 unit increments is assigned. Participants with EDSS scores of 0.0 to 4.5 are fully ambulatory; patients with EDSS scores of 5.0 to 9.5 have impaired ambulation.
  units on a scale | 2.62 (1.138) | 2.65 (1.135) | 2.61 (1.160) | 2.62 (1.144)
Time Since MS Symptom Onset [Mean (Standard Deviation); unit: years] | 6.88 (5.877) | 7.16 (6.255) | 6.85 (6.449) | 6.96 (6.195)
Time Since MS Diagnosis [Mean (Standard Deviation); unit: years] | 3.71 (4.361) | 3.70 (4.518) | 3.60 (4.193) | 3.67 (4.357)
Age at MS Symptom Onset [Mean (Standard Deviation); unit: years] | 29.5 (8.92) | 29.3 (9.25) | 28.4 (8.42) | 29.1 (8.88)
Age at MS Diagnosis [Mean (Standard Deviation); unit: years] | 32.7 (9.01) | 32.7 (9.49) | 31.6 (8.81) | 32.4 (9.12)

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Annualized Relapse Rate (ARR) During the Treatment Period
Description: The relapse rate was based on confirmed relapses. A relapse was defined as new or worsening neurological symptoms attributable to MS and preceded by a relatively stable or improving neurological state for at least 30 days. Symptoms must have persisted for > 24 hours and not be attributable to confounding clinical factors. Relapses were confirmed when accompanied by objective neurological worsening based on examination by the blinded evaluator, consistent with an increase of ≥ 0.5 on the overall EDSS score relative to the most recent EDSS assessment, or 2 points on one of the functional system scale scores, or 1 point on ≥ two functional system scale scores.
  Relapse rate was calculated as the total number of relapses divided by the total number of days in the study * 365.25.
  ARR was adjusted for region (Eastern Europe vs rest of world), Baseline age, and Baseline number of gadolinium-enhancing lesions; the natural log transformation of time on study was included as an offset term.
Time Frame: 12 months
Population: The ITT population consisted of all randomized participants who received at least 1 dose of study medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: relapses/year
Arm/Group | Interferon Beta-1a | Ozanimod 0.5 mg | Ozanimod 1 mg
Number analyzed (Participants) | 448 | 451 | 447
relapses/year | 0.350 [0.279 to 0.440] | 0.241 [0.188 to 0.308] | 0.181 [0.140 to 0.236]
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Ozanimod 1 mg; Test type: Superiority; p < 0.0001, Poisson regression model — To account for multiple comparisons, each of the 2 treatment comparisons was tested at the alpha = 0.025 level; Adjusted for region, Baseline age, number of gadolinium enhancing (GdE) lesions and included the natural log transformation of time as an offset term; Rate Ratio = 0.518, 95% CI 2-sided [0.405 to 0.663]
Statistical Analysis 2: Comparison: Interferon Beta-1a vs Ozanimod 0.5 mg; Test type: Superiority; p = 0.0013, Poisson Regression Model — To account for multiple comparisons, each of the 2 treatment comparisons was tested at the alpha = 0.025 level; Adjusted for region, Baseline age and the number of GdE lesions, and included the natural log transformation of time on study as an offset term; Rate Ratio = 0.688, 95% CI 2-sided [0.547 to 0.864]

2. Secondary Outcome: Adjusted Mean Number of New or Enlarging Hyperintense T2-Weighted Brain Magnetic Resonance Imaging (MRI) Lesions Per Scan Over 12 Months
Description: The number of new or enlarging hyperintense T2-weighted brain MRI lesions per scan was based on the cumulative number of new or enlarging T2 lesions since Baseline over treatment period.
Time Frame: 12 month treatment period; MRI scans were assessed at Month 6 and Month 12
Population: ITT population; participants with non-missing MRI results.
Measure: Least Squares Mean (95% Confidence Interval); unit: T2 lesions/scan
Arm/Group | Interferon Beta-1a | Ozanimod 0.5 mg | Ozanimod 1 mg
Number analyzed (Participants) | 382 | 397 | 388
T2 lesions/scan | 2.836 [2.331 to 3.451] | 2.139 [1.777 to 2.575] | 1.465 [1.203 to 1.784]
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Ozanimod 1 mg; Test type: Superiority; p < 0.0001, Negative Binomial Regression Model — To account for multiple comparisons, each of the 2 treatment comparisons was tested at the alpha = 0.05 level; Adjusted for region, Baseline age and GdE lesions; included the natural log transformation of available MRI scans over 12 months as an offset term; Rate Ratio = 0.517, 95% CI 2-sided [0.427 to 0.625] — Rate Ratio = Ozanimod / IFN β-1a
Statistical Analysis 2: Comparison: Interferon Beta-1a vs Ozanimod 0.5 mg; Test type: Superiority; p = 0.0032, Negative binomial regression model — To account for multiple comparisons, each of the 2 treatment comparisons was tested at the alpha = 0.05 level; [statistical method as in outcome 2, analysis 1]; Rate Ratio = 0.754, 95% CI 2-sided [0.625 to 0.910] — Rate Ratio = Ozanimod / IFN β-1a

3. Secondary Outcome: Adjusted Mean Number of Gadolinium Enhancing (GdE) Brain MRI Lesions at Month 12
Time Frame: Month 12
Population: ITT population; participants with non-missing MRI results.
Measure: Least Squares Mean (95% Confidence Interval); unit: lesions
Arm/Group | Interferon Beta-1a | Ozanimod 0.5 mg | Ozanimod 1 mg
Number analyzed (Participants) | 382 | 397 | 388
lesions | 0.433 [0.295 to 0.635] | 0.287 [0.197 to 0.418] | 0.160 [0.106 to 0.242]
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Ozanimod 1 mg; Test type: Superiority; p < 0.0001, Negative Binomial Regression Model — To account for multiple comparisons, each of the 2 treatment comparisons was tested at the alpha = 0.05 level; Adjusted for region, Baseline age and GdE lesions; included the natural log transformation of available MRI scans as an offset term; Rate Ratio = 0.370, 95% CI 2-sided [0.256 to 0.536]
Statistical Analysis 2: Comparison: Interferon Beta-1a vs Ozanimod 0.5 mg; Test type: Superiority; p = 0.0182, Negative binomial regression model — To account for multiple comparisons, each of the 2 treatment comparisons was tested at the alpha = 0.05 level; [statistical method as in outcome 3, analysis 1]; Rate Ratio = 0.662, 95% CI 2-sided [0.471 to 0.932]

4. Secondary Outcome: Time to Onset of Disability Progression Confirmed After 3 Months
Description: EDSS is used to quantify disability and disability progression over time in MS. Based on a neurological examination, 8 functional systems (visual, brain stem, pyramidal, cerebellar, sensory, bowel & bladder, cerebral, and other functions) are scored from 0 (no disability) to 5 or 6 (more severe disability). Ambulation is assessed based on distance the patient is able to walk, whether assistance is required or restrictions are present.
  The EDSS score ranges from 0 (normal) to 10 (death due to MS) in 0.5 unit increments.
  Disability progression is defined by a sustained worsening in EDSS score of 1.0 point or more confirmed after 3 months. Time to onset of disability progression was calculated from the date of first dose to the date of the first visit at which the 1.0 point increase in EDSS was met using Kaplan-Meier methods. Participants without a sustained disease progression event were censored on the date of their last assessment or last dose of study drug, whichever was later.
Time Frame: From first dose to the end of the 12-month treatment period
Population: ITT population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Interferon Beta-1a | Ozanimod 0.5 mg | Ozanimod 1 mg
Number analyzed (Participants) | 448 | 451 | 447
days | NA [NA to NA] — Not estimable as there were insufficient disability events | NA [NA to NA] — Not estimable as there were insufficient disability events | NA [NA to NA] — Not estimable as there were insufficient disability events
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Ozanimod 1 mg; Test type: Superiority; p = 0.3055, Cox proportional hazards model; Based on the Cox proportional hazard model with factors for treatment group, adjusted for region, Baseline age, and Baseline EDSS score; Hazard Ratio (HR) = 0.690, 95% CI 2-sided [0.340 to 1.402] — Hazard Ratio (Ozanimod / IFN β-1a)
Statistical Analysis 2: Comparison: Interferon Beta-1a vs Ozanimod 0.5 mg; Test type: Superiority; p = 0.7163, Cox proportional hazards model; Based on the Cox proportional hazard model with factors for treatment group, adjusted for region, Baseline age and Baseline EDSS score; Hazard Ratio (HR) = 0.886, 95% CI 2-sided [0.460 to 1.705] — Hazard Ratio (Ozanimod / IFN β-1a)

5. Secondary Outcome: Time to Onset of Disability Progression Confirmed After 6 Months
Description: EDSS is used to quantify disability and disability progression over time in MS. Based on a neurological examination, 8 functional systems (visual, brain stem, pyramidal, cerebellar, sensory, bowel & bladder, cerebral, and other functions) are scored from 0 (no disability) to 5 or 6 (more severe disability). Ambulation is assessed based on distance the patient is able to walk, whether assistance is required or restrictions are present.
  The EDSS score ranges from 0 (normal) to 10 (death due to MS) in 0.5 unit increments.
  Disability progression is defined by a sustained worsening in EDSS score of 1.0 point or more confirmed after 6 months. Time to onset of disability progression was calculated from the date of first dose to the date of the first visit at which the 1.0 point increase in EDSS was met using Kaplan-Meier methods. Participants without a sustained disease progression event were censored on the date of their last assessment or last dose of study drug, whichever was later.
Time Frame: From first dose to the end of the 12-month treatment period
Population: ITT population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Interferon Beta-1a | Ozanimod 0.5 mg | Ozanimod 1 mg
Number analyzed (Participants) | 448 | 451 | 447
days | NA [NA to NA] — Not estimable as there were insufficient disability events | NA [NA to NA] — Not estimable as there were insufficient disability events | NA [NA to NA] — Not estimable as there were insufficient disability events
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Ozanimod 1 mg; Test type: Superiority; p = 0.6725, Cox proportional hazards model; [statistical method as in outcome 4, analysis 2]; Hazard Ratio (HR) = 1.238, 95% CI 2-sided [0.460 to 3.337] — Hazard Ratio (Ozanimod / IFN β-1a)
Statistical Analysis 2: Comparison: Interferon Beta-1a vs Ozanimod 0.5 mg; Test type: Superiority; p = 0.3755, Cox proportional hazard model; [statistical method as in outcome 4, analysis 2]; Hazard Ratio (HR) = 1.535, 95% CI 2-sided [0.595 to 3.963] — Hazard Ratio (Ozanimod / IFN β-1a)

6. Secondary Outcome: Percentage of Participants Who Were Gadolinium Enhancing Lesion-Free at Month 12
Description: MRI scans were analyzed by blinded centralized reading facility.
Time Frame: Month 12
Population: The ITT population; Participants who were missing the Month 12 MRI data were considered non-responders; ie, as not being lesion-free (non-responder imputation).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Interferon Beta-1a | Ozanimod 0.5 mg | Ozanimod 1 mg
Number analyzed (Participants) | 448 | 451 | 447
percentage of participants | 63.17 [58.70 to 67.64] | 68.29 [64.00 to 72.59] | 74.05 [69.99 to 78.11]
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Ozanimod 1 mg; Test type: Superiority; p = 0.0006, Cochran-Mantel-Haenszel; Based on the CMH test stratified by region and EDSS category per Interactive Voice Response System (IVRS); Difference in Percentages = 10.88, 95% CI 2-sided [4.84 to 16.92]
Statistical Analysis 2: Comparison: Interferon Beta-1a vs Ozanimod 0.5 mg; Test type: Superiority; p = 0.1130, Cochran-Mantel-Haenszel; Based on the CMH test stratified by region and EDSS category per IVRS; Difference in Percentages = 5.12, 95% CI 2-sided [-1.07 to 11.32]

7. Secondary Outcome: Percentage of Participants Who Were T2 Lesion-Free at Month 12
Description: MRI scans were analyzed by blinded centralized reading facility.
Time Frame: Month 12
Population: The ITT population; participants who were missing the Month 12 MRI data were considered non-responders, ie, as not being lesion-free.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Interferon Beta-1a | Ozanimod 0.5 mg | Ozanimod 1 mg
Number analyzed (Participants) | 448 | 451 | 447
percentage of participants | 23.44 [19.51 to 27.36] | 26.39 [22.32 to 30.45] | 27.96 [23.80 to 32.12]
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Ozanimod 1 mg; Test type: Superiority; p = 0.1180, Cochran-Mantel-Haenszel; Based on the CMH test stratified by region and EDSS Scale category per IVRS; Difference in Percentages = 4.53, 95% CI 2-sided [-1.19 to 10.24]
Statistical Analysis 2: Comparison: Interferon Beta-1a vs Ozanimod 0.5 mg; Test type: Superiority; p = 0.3023, Cochran-Mantel-Haenszel; Based on the CMH test stratified by region and EDSS Scale category per IVRS; Difference in percentages = 2.95, 95% CI 2-sided [-2.70 to 8.60]

8. Secondary Outcome: Percent Change From Baseline in Normalized Brain Volume at Month 12
Description: Brain volume (a measure of brain atrophy) was analyzed by MRI.
Time Frame: Baseline to Month 12
Population: The ITT population with available MRI data at Baseline and Month 12
Measure: Median (Full Range); unit: percent change
Arm/Group | Interferon Beta-1a | Ozanimod 0.5 mg | Ozanimod 1 mg
Number analyzed (Participants) | 334 | 347 | 338
percent change | -0.57 [-3.7 to 1.1] | -0.50 [-2.7 to 1.4] | -0.39 [-2.8 to 2.1]
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Ozanimod 1 mg; Due to the non-normal distribution of the data for brain volume loss, the analyses for percent change from baseline in normalized brain volume were compared using rank-ANCOVA, adjusted for region (Eastern Europe vs Rest of World), and EDSS category per IVRS, with the dependent variable as the residual of the rank of brain volume at Baseline regressed on rank of percent change; Test type: Superiority; p < 0.0001, Rank ANCOVA; Adjusted for region and EDSS category per IVRS
Statistical Analysis 2: Comparison: Interferon Beta-1a vs Ozanimod 0.5 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0615, Rank ANCOVA; Adjusted for region and EDSS Scale per IVRS

9. Secondary Outcome: Change From Baseline to Month 12 in Multiple Sclerosis Functional Composite (MSFC) Score Including the Low-Contrast Letter Acuity (LCLA) Test
Description: The MSFC-LCLA is a battery including the following 4 individual scales:
  * Timed 25-Foot Walk is an ambulation measure of walking 25 feet with time taken recorded in seconds
  * 9-Hole Peg Test (9HPT) is a quantitative measure of upper extremity (arm and hand) function
  * Symbol Digit Modalities Test (SDMT) is a measure of executive cognitive function that assesses processing speed, flexibility, and calculation ability
  * Low-Contrast Letter Acuity Test (LCLA) used a standardized set of charts to assess low contrast visual acuity, charts are scored according to the number of letters that are identified correctly
  Z-scores were calculated for for each component and averaged to create an overall composite score, using the study population as the reference population. A z-score represents the number of standard deviations a patient's test result is higher (z > 0) or lower (z < 0) than the average test result (z = 0) of the reference population. A positive change indicates improvement.
Time Frame: Baseline to Month 12
Population: The ITT population with available Baseline and Month 12 MSFC z-scores.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Interferon Beta-1a | Ozanimod 0.5 mg | Ozanimod 1 mg
Number analyzed (Participants) | 447 | 450 | 447
z-score | -0.022 (0.334) | -0.007 (0.351) | 0.003 (0.328)
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Ozanimod 1 mg; Test type: Superiority; p = 0.1290, ANCOVA; Adjusted for region, EDSS category per IVRS and the Baseline MSFC score; LS Mean Difference = 0.034, 95% CI 2-sided [-0.010 to 0.077]
Statistical Analysis 2: Comparison: Interferon Beta-1a vs Ozanimod 0.5 mg; Test type: Superiority; p = 0.4942, ANCOVA; Adjusted for region, EDSS category per IVRS and the Baseline MSFC score; LS Mean Difference = 0.015, 95% CI 2-sided [-0.028 to 0.059]

10. Secondary Outcome: Mean Change From Baseline in Multiple Sclerosis Quality of Life (MSQOL)-54 Physical Health Composite Summary and Mental Health Composite Summary Scores
Description: The MSQOL-54 is a multidimensional health-related QOL measure that combines both generic and MS-specific items into a single instrument. The instrument includes 12 subscales, two summary scores, and two single-item measures.
  The two summary scores - physical health and mental health - are derived from a weighted combination of scale scores.
  The physical health composite score includes Physical function, Health perceptions, Energy/fatigue, Role limitations - physical, Pain, Sexual function, Social function, and Health distress.
  The mental health composite score includes Health distress, Overall quality of life, Emotional well-being, Role limitations - emotional, and Cognitive function.
  Each composite summary score has a range from 0 to 100 where higher scores indicate better quality of life. A positive change from Baseline indicates improvement.
Time Frame: Baseline to Month 12
Population: ITT population with available Baseline data; missing post-baseline data were imputed using a mixed-effects regression model (random slope and intercept).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interferon Beta-1a | Ozanimod 0.5 mg | Ozanimod 1 mg
Number analyzed (Participants) | 448 | 451 | 446
units on a scale
  Physical health composite summary: number analyzed (Participants) | 445 | 448 | 443
  Physical health composite summary | 0.046 (12.578) | 1.414 (12.343) | 1.925 (11.870)
  Mental health composite summary | -0.123 (15.240) | 0.283 (15.686) | 0.260 (15.800)
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Ozanimod 1 mg; Analysis of Physical Health Composite Summary; Test type: Superiority; p = 0.0364, ANCOVA; Adjusted for region, EDSS category per IVRS, and the Baseline summary score; Mean Difference (Final Values) = 1.642, 95% CI 2-sided [0.104 to 3.180]
Statistical Analysis 2: Comparison: Interferon Beta-1a vs Ozanimod 0.5 mg; Analysis of Physical Health Composite Summary; Test type: Superiority; p = 0.1905, ANCOVA; Adjusted for region, EDSS category per IVRS, and the Baseline summary score; Mean Difference (Final Values) = 1.024, 95% CI 2-sided [-0.510 to 2.559]
Statistical Analysis 3: Comparison: Interferon Beta-1a vs Ozanimod 1 mg; Analysis of Mental Health Composite Summary; Test type: Superiority; p = 0.7104, ANCOVA; Adjusted for region, EDSS category per IVRS, and the Baseline summary score; Mean Difference (Final Values) = 0.356, 95% CI 2-sided [-1.523 to 2.234]
Statistical Analysis 4: Comparison: Interferon Beta-1a vs Ozanimod 0.5 mg; Analysis of Mental Health Composite Summary; Test type: Superiority; p = 0.8587, ANCOVA; Adjusted for region, EDSS category per IVRS, and the Baseline summary score; Mean Difference (Final Values) = -0.170, 95% CI 2-sided [-2.045 to 1.705]

11. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence that does not necessarily have a causal relationship with the investigational product (IP). An AE can be any unfavorable or unintended sign, including an abnormal laboratory finding, symptom or disease temporally associated with the use of an IP whether or not considered related to the IP. A serious AE (SAE) is any untoward medical occurrence or effect that results in death, is life-threatening, requires hospitalization or prolongation of existing inpatient hospitalization. The investigator assessed the severity of AEs as mild, moderate, or severe.
Time Frame: From the first dose of study drug until 28 days following the last dose of study drug; mean exposure to study drug was 13.5 months for interferon beta-1a and 13.6 months for each ozanimod group.
Population: Safety Population consisted of all participants who received at least 1 dose of randomized study medication, analyzed according to the highest dose of ozanimod treatment actually received (up to 1 mg) and not according to the treatment they were randomized to receive, if different.
Measure: Count of Participants; unit: Participants
Groups:
- Ozanimod 1 mg: Participants received ozanimod 0.5 mg orally once a day and a placebo intramuscular injection weekly until the last participant had been treated for at least 12 months.
Arm/Group | Interferon Beta-1a | Ozanimod 0.5 mg | Ozanimod 1 mg
Number analyzed (Participants) | 445 | 453 | 448
Participants
  Any TEAE | 336 | 259 | 268
  Any Moderate or Severe TEAE | 182 | 113 | 138
  Any Severe TEAE | 10 | 10 | 7
  Any Suspected TEAE | 83 | 76 | 91
  Any Related TEAE | 13 | 8 | 7
  Any Serious TEAE | 11 | 16 | 13
  Any Suspected Serious TEAE | 0 | 0 | 3
  Any Related Serious TEAE | 0 | 0 | 1
  Any TEAE Leading to Stopping of Study Drug | 16 | 7 | 13
  Any TEAE Leading to Study Withdrawal | 16 | 7 | 13
  Any Death | 0 | 0 | 0
  Any Death related to Study Drug | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study drug until 28 days following the last dose of study drug; mean exposure to study drug was 13.5 months for interferon beta-1a and 13.6 months for each ozanimod group.
Description: The Safety population included all participants who received at least 1 dose of randomized study drug. All participants in the Safety population were analyzed according to the highest dose of ozanimod treatment actually received (up to 1 mg) and not according to the treatment they were randomized to receive, if different.
Arm/Group | Interferon Beta-1a | Ozanimod 0.5 mg | Ozanimod 1 mg
Serious Adverse Events (participants affected / at risk) | 11/445 | 16/453 | 13/448
Other Adverse Events (participants affected / at risk) | 273/445 | 88/453 | 57/448
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Interferon Beta-1a (N=445) | Ozanimod 0.5 mg (N=453) | Ozanimod 1 mg (N=448)
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 0
Sinus Bradycardia (Cardiac disorders) | 0 | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 0 | 0 | 1
Duodenal Ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Gallbladder Polyp (Hepatobiliary disorders) | 0 | 1 | 0
Appendiceal Abscess (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0
Lyme Disease (Infections and infestations) | 1 | 0 | 0
Postoperative Abscess (Infections and infestations) | 0 | 0 | 1
Pyelonephritis Acute (Infections and infestations) | 1 | 0 | 1
Subcutaneous Abscess (Infections and infestations) | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Eye Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fibrin D Dimer Increased (Investigations) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Benign Ovarian Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Fibroadenoma Of Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Invasive Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Testicular Seminoma (Pure) Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebral Infarction (Nervous system disorders) | 1 | 0 | 0
Cervical Radiculopathy (Nervous system disorders) | 0 | 1 | 0
Multiple Sclerosis Relapse (Nervous system disorders) | 2 | 0 | 0
Myelopathy (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Vascular Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Renal Colic (Renal and urinary disorders) | 0 | 1 | 1
Menometrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Postmenopausal Haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Interferon Beta-1a (N=445) | Ozanimod 0.5 mg (N=453) | Ozanimod 1 mg (N=448)
Influenza Like Illness (General disorders) | 227 | 18 | 17
Pyrexia (General disorders) | 28 | 5 | 5
Nasopharyngitis (Infections and infestations) | 36 | 44 | 30
Upper Respiratory Tract Infection (Infections and infestations) | 24 | 31 | 18
Headache (Nervous system disorders) | 25 | 27 | 34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than one (1) year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene sixty (60) days prior to submission. Celgene may remove confidential and/or proprietary information before publication